CLINICAL TRIAL: NCT02468921
Title: The Impact of Surgical Treatment of Benign Non-toxic Goiter on the Voice Function
Brief Title: Goitres Influence on Voice Function - The Impact of Surgery
Acronym: SOLOIST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Roed Sorensen, MD, University of Southern Denmark
Other Study IDs: S-20131
Record Dates: First submitted 2015-01-19; First posted 2015-06-11 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Goiter
Keywords: Goitre; thyroid disease; struma
MeSH Terms: conditions — Goiter; Thyroid Diseases | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Thyroidectomy — Regular thyroidectomy or hemithyroidectomy through Kocher's skin incision

SUMMARY:
The aim of the study is to investigate the influence benign non-toxic goitre and the surgical treatment hereof on the voice function before and 6 months following surgery.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing hemi- or total thyroidectomy for benign non-toxic goiter with pressure symptoms
* The patients must be able to understand, write and read Danish

Exclusion criteria:

* Previous surgery to the neck
* Diabetes or any neuromuscular disorders.
* Present or previous head and neck malignancy, including malignancy found in the surgical thyroid specimen or suspicion hereof.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing hemi- or total thyroidectomy at Odense University Hospital for benign symptomatic non-toxic goiter
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with changed frequency range in voice function following thyroidectomy | 6 months
  Change in frequency range (Hz) of the Voice Range Profiler Phonetogram from baseline to 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Godballe, Professor, Study Director — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark